CLINICAL TRIAL: NCT03117868
Title: Mortality of Patients Undergoing Fracture of the Upper Extremity u Femur at the University Hospital of Amiens
Acronym: FESF-Amiens
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-04
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Femur Fracture; Morality
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study of mortality at 6 months — The objective is to provide strong arguments for establishing a dynamic of collective care for patients suffering from an EFSF

SUMMARY:
Fractures of the upper femur (EFSF) represent a major public health problem in the elderly. Approximately 1.6 million patients are victims each year of an EFSF and this number is increasing as a result of the aging of the population.

In a recent Amiens retrospective study the mortality was estimated to be 22.5% at 1 year of the fracture. In surviving patients, the impact on loss of autonomy and degradation of quality of life is considerable.

The reduction of the incidence of post-operative complications includes the identification of risk factors.

No prospective study in Amiens has investigated the mortality and the study of the variables involved in the prognosis and long-term mortality of these patients.

ELIGIBILITY:
Inclusion Criteria:

* All the patients operated from a fracture of traumatic origin of the ESF to the emergency block at the CHU of Amiens
* Patients transferred to the CHU after being cared for in another structure will be included.
* If a patient successively presents a fracture of each upper extremity of the femur outside of a surgical resumption, two inclusions will be realized

Exclusion Criteria:

* Do not include non-traumatic fractures of the upper end of the femur (pathological fractures: cancer, for example)
* Fractures of the upper end of the femur associated with polytrauma will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients operated with an EFSF and meeting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Mortality at 6 months of EFSF patients | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France